CLINICAL TRIAL: NCT04608305
Title: A Phase I/II Randomized, Multi-Center, Placebo-Controlled, Dose-Escalation Study to Evaluate the Safety, Immunogenicity and Potential Efficacy of an rVSV-SARS-CoV-2-S Vaccine (IIBR-100) in Adults
Brief Title: Evaluate the Safety, Immunogenicity and Potential Efficacy of an rVSV-SARS-CoV-2-S Vaccine
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Israel Institute for Biological Research (IIBR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IIBR 20-001
Record Dates: First submitted 2020-10-26; First posted 2020-10-29 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Covid19
Keywords: SARS-CoV-2; Vaccine
MeSH Terms: conditions — COVID-19 | interventions — rVSV-deltaG-spike COVID-19 vaccine; PRIME protocol; Single Person

STUDY DESIGN:
Intervention Model Description: The study is comprised of two phases, a dose-escalation Phase I (sentinels + expansions) and expansion to Phase II that includes larger cohorts, elderly age groups and additional boost injection. Subjects will be randomly allocated to the study groups in both phases.
  Dosing of prime during phase I occurred in a sequential fashion (partially overlapping), starting from low-dose and continuing to mid and high doses following safety reviews. Prior to expansion to phase II, cumulative data from phase I was evaluated (dose and regimen) by the data safety monitoring board. The DSMB's recommendations regarding expansion to phase II were the continuation of prime-boost regimens of medium, high and top doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (18):
- phase I - Group Ia, prime, low dose (Experimental): Male and female subjects (18-55 years old) administered with a single-dose of IIBR-100 1*10E5 pfu/ml or saline placebo at day 0
  Interventions: Biological: IIBR-100, low dose (prime); Other: Saline Placebo (single)
- phase I - Group Ib, Prime, medium dose (Experimental): Male and female subjects (18-55 years old) administered with a single-dose of IIBR-100 1*10E6 pfu/ml or saline placebo at day 0
  Interventions: Biological: IIBR-100 medium dose (prime); Other: Saline Placebo (single)
- phase I - Group Ic, Prime, high dose (Experimental): Male and female subjects (18-55 years old) administered with a single-dose of IIBR-100 1*10E7 pfu/ml or saline placebo at day 0
  Interventions: Biological: IIBR-100 high-dose (prime); Other: Saline Placebo (single)
- phase I - Group Id, prime-boost, low dose (Experimental): Male and female subjects (18-55 years old) administered twice with IIBR-100 1*10E5 pfu/ml or saline placebo, 4 weeks apart, at days 0 and 28.
  Interventions: Biological: IIBR-100 low-dose (prime-boost); Other: Saline Placebo (double)
- phase II - Group IIa, prime, low dose* (Experimental): Male and female subjects (18-55 years old) administered with a single-dose of IIBR-100 1*10E5 pfu/ml or saline placebo at day 0.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100, low dose (prime); Other: Saline Placebo (single)
- Phase II - Group IIb, Prime, low dose, elderly subjects* (Experimental): Male and female subjects (56-85 years old) administered with a single-dose of IIBR-100 1*10E5 pfu/ml or saline placebo at day 0.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100, low dose (prime); Other: Saline Placebo (single)
- phase II - Group IIc, Prime, medium dose* (Experimental): Male and female subjects (18-55 years old) administered with a single-dose of IIBR-100 1*10E6 pfu/ml or saline placebo at day 0.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100 medium dose (prime); Other: Saline Placebo (single)
- phase II - Group IId, Prime, medium dose, elderly subjects* (Experimental): Male and female subjects (56-85 years old) administered with a single-dose of IIBR-100 1*10E6 pfu/ml or saline placebo at day 0.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100 medium dose (prime); Other: Saline Placebo (single)
- Phase II - Group IIe, prime, high dose* (Experimental): Male and female subjects (18-55 years old) administered with a single-dose of IIBR-100 1*10E7 pfu/ml or saline placebo at day 0.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100 high-dose (prime); Other: Saline Placebo (single)
- Phase II - Group IIf, Prime, high dose, elderly subjects* (Experimental): Male and female subjects (56-85 years old) administered with a single-dose of IIBR-100 1*10E7 pfu/ml or saline placebo at day 0.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100 high-dose (prime); Other: Saline Placebo (single)
- phase II - Group IIg, prime-boost, low dose* (Experimental): Male and female subjects (18-55 years old) administered twice with IIBR-100 1*10E5 pfu/ml or saline placebo, 4 weeks apart at days 0 and 28.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100 low-dose (prime-boost); Other: Saline Placebo (double)
- phase II - Group IIh, prime-boost, low dose, elderly subjects* (Experimental): Male and female subjects (56-85 years old) administered twice with IIBR-100 1*10E5 pfu/ml or saline placebo, 4 weeks apart, at days 0 and 28.
  *Treatment arm was deactivated based on immunogenicity data and DSMB recommendations.
  Interventions: Biological: IIBR-100 low-dose (prime-boost); Other: Saline Placebo (double)
- phase II - Group IIi, prime-boost, medium dose (Experimental): Male and female subjects (18-55 years old) administered twice with IIBR-100 1*10E6 pfu/ml or saline placebo, 4 weeks apart at days 0 and 28.
  Interventions: Other: Saline Placebo (double); Biological: IIBR-100 medium-dose (prime-boost)
- phase II - Group IIj, prime-boost, medium dose, elderly subjects (Experimental): Male and female subjects (56-85 years old) administered twice with IIBR-100 1*10E6 pfu/ml or saline placebo, 4 weeks apart, at days 0 and 28.
  Interventions: Other: Saline Placebo (double); Biological: IIBR-100 medium-dose (prime-boost)
- phase II - Group IIk, prime-boost, high dose (Experimental): Male and female subjects (18-55 years old) administered twice with IIBR-100 1*10E7 pfu/ml or saline placebo, 4 weeks apart at days 0 and 28.
  Interventions: Other: Saline Placebo (double); Biological: IIBR-100 high-dose (prime-boost)
- phase II - Group IIl, prime-boost, high dose, elderly subjects (Experimental): Male and female subjects (56-85 years old) administered twice with IIBR-100 1*10E7 pfu/ml or saline placebo, 4 weeks apart, at days 0 and 28.
  Interventions: Other: Saline Placebo (double); Biological: IIBR-100 high-dose (prime-boost)
- phase II - Group IIm, prime-boost, top dose (Experimental): Male and female subjects (18-55 years old) administered twice with IIBR-100 1*10E8 pfu/ml or saline placebo, 4 weeks apart at days 0 and 28.
  Interventions: Other: Saline Placebo (double); Biological: IIBR-100 top-dose (prime-boost)
- phase II - Group IIn, prime-boost, top dose, elderly subjects (Experimental): Male and female subjects (56-85 years old) administered twice with IIBR-100 1*10E8 pfu/ml or saline placebo, 4 weeks apart, at days 0 and 28.
  Interventions: Other: Saline Placebo (double); Biological: IIBR-100 top-dose (prime-boost)

INTERVENTIONS:
Biological: IIBR-100, low dose (prime) — Single administration of IIBR-100 1*10E5 pfu/ml
  Arms: Phase II - Group IIb, Prime, low dose, elderly subjects*; phase I - Group Ia, prime, low dose; phase II - Group IIa, prime, low dose*
Biological: IIBR-100 medium dose (prime) — Single administration of IIBR-100 1*10E6 pfu/ml
  Arms: phase I - Group Ib, Prime, medium dose; phase II - Group IIc, Prime, medium dose*; phase II - Group IId, Prime, medium dose, elderly subjects*
Biological: IIBR-100 high-dose (prime) — Single administration of IIBR-100 1*10E7 pfu/ml
  Arms: Phase II - Group IIe, prime, high dose*; Phase II - Group IIf, Prime, high dose, elderly subjects*; phase I - Group Ic, Prime, high dose
Biological: IIBR-100 low-dose (prime-boost) — Two administrations of IIBR-100 1*10E5 pfu/ml, 28 days apart
  Arms: phase I - Group Id, prime-boost, low dose; phase II - Group IIg, prime-boost, low dose*; phase II - Group IIh, prime-boost, low dose, elderly subjects*
Other: Saline Placebo (single) — Single administration of saline placebo
  Arms: Phase II - Group IIb, Prime, low dose, elderly subjects*; Phase II - Group IIe, prime, high dose*; Phase II - Group IIf, Prime, high dose, elderly subjects*; phase I - Group Ia, prime, low dose; phase I - Group Ib, Prime, medium dose; phase I - Group Ic, Prime, high dose; phase II - Group IIa, prime, low dose*; phase II - Group IIc, Prime, medium dose*; phase II - Group IId, Prime, medium dose, elderly subjects*
Other: Saline Placebo (double) — Two administrations of saline placebo, 28 days apart
  Arms: phase I - Group Id, prime-boost, low dose; phase II - Group IIg, prime-boost, low dose*; phase II - Group IIh, prime-boost, low dose, elderly subjects*; phase II - Group IIi, prime-boost, medium dose; phase II - Group IIj, prime-boost, medium dose, elderly subjects; phase II - Group IIk, prime-boost, high dose; phase II - Group IIl, prime-boost, high dose, elderly subjects; phase II - Group IIm, prime-boost, top dose; phase II - Group IIn, prime-boost, top dose, elderly subjects
Biological: IIBR-100 medium-dose (prime-boost) — Two administrations of IIBR-100 1*10E6 pfu/ml, 28 days apart
  Arms: phase II - Group IIi, prime-boost, medium dose; phase II - Group IIj, prime-boost, medium dose, elderly subjects
Biological: IIBR-100 high-dose (prime-boost) — Two administrations of IIBR-100 1*10E7 pfu/ml, 28 days apart
  Arms: phase II - Group IIk, prime-boost, high dose; phase II - Group IIl, prime-boost, high dose, elderly subjects
Biological: IIBR-100 top-dose (prime-boost) — Two administrations of IIBR-100 1*10E8 pfu/ml, 28 days apart
  Arms: phase II - Group IIm, prime-boost, top dose; phase II - Group IIn, prime-boost, top dose, elderly subjects

SUMMARY:
The SARS-CoV-2 virus is responsible for the COVID-19 pandemic. The pandemic emerged from Wuhan Province in China in December 2019 and was declared by the WHO Director-General a Public Health Emergency of International Concern on 30 January 2020.

In this study, a vaccine developed by IIBR for SARS-CoV-2 virus will be assessed for its safety and potential efficacy in volunteers. The study is comprised of two phases, a dose-escalation phase (phase I) during which subjects (18-55 years old) will be randomly allocated to receive a single administration of IIBR-100 at low, mid or high dose or saline or two administrations of IIBR-100 at low dose, or saline, 28 days apart.

Based on results obtained during phase I, and cumulative phase I data review, the expansion phase (phase II) has begun, during which larger cohorts as well as elderly age subjects were initially planned to be randomly allocated to receive a single administration of IIBR-100 at low, mid or high dose or saline, or two administrations of IIBR-100 at low, mid or high dose (prime-boost) or saline, 28 days apart. Additional top-dose (prime-boost) may be implemented when immunogenicity of any prime-boost arm is considered insufficient. However, based on immunogenicity preliminary data and DSMB recommendations, only the two administrations of mid, high and top dose (prime-boost) or saline will continue in the study.

The subjects will be followed for a period of up to 12 months post last vaccine administration to assess the safety and efficacy of the vaccine.

DETAILED DESCRIPTION:
In the Phase I, healthy adult volunteers will be randomly allocated to one of the four treatment groups to receive a single administration (prime) of IIBR-100 at low, mid or high dose or saline or two administrations (prime-boost) of IIBR-100 at low dose, or saline, 28 days apart. During Phase I, dosing of prime will proceed in a sequential fashion followed by a safety review committee and DSMB to consider expansion to include the rest of the group and escalation to the next groups. Only Groups that demonstrate acceptable safety profile, immunogenicity and potential efficacy will be included in the Phase II operation. In both phases, the subjects will receive an intramuscular injection of the IIBR-100 consisted of 1ml replicating viral rVSV SARS-CoV-2-S vaccine or placebo consisted of 1ml of 0.9% saline. Dosing will be performed at Day 0 and Day 28 (for allocated to prime-boost treatment groups) in the deltoid muscle and will be followed through 12 months post last vaccination. Follow-up visits for subjects administered with the single administration (prime) or placebo will occur at 1, 2 and 4 weeks as well as 2, 3, 6, 9 and 12 months after dosing. Follow up visits for subjects administered with two administrations (prime-boost) or placebo will occur at 1, 2 and 4 weeks post each vaccination as well as at 2, 3, 6, 9 and 12 months after the second vaccination. Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions from the time of each dosing through 7 days post each dosing. Unsolicited non-serious safety events will be collected from the time of each dosing through 28 days post each dosing. Serious safety events, new-onset chronic medical conditions and medically attended safety events will be collected through 12 months after the last dosing.

ELIGIBILITY:
Inclusion Criteria:

Phase I (abbreviated):

* Healthy males or females, ages 18 to 55 (inclusive) at the time of screening.
* Negative PCR and no presence of ELISA antibody titers to SARS-CoV-2 at screening.
* Females of childbearing potential and males must be willing to use effective methods of contraception such as hormones (OCP, oral contraceptive pill), condom or occlusive cap with spermicidal agents, intrauterine device (IUD) or intrauterine system (IUS) from at least 14 days prior to vaccination through 90 days following last injection.
* Subjects in general good health with no chronic disease nor consumes chronic medication in the opinion of the investigator as determined by medical history, vital signs and a physical examination.
* No clinically significant abnormalities in hematology, blood chemistry, or urinalysis laboratory tests at screening.
* Negative HIV, Hepatitis B and Hepatitis C serology tests.
* Normal oral temperature, normal sinus rhythm, pulse rate no greater than 100 beats per minute and normal systolic blood pressure (below 140/90 mmHg)
* Must be willing to forgo blood donation during the blood drawing phase of the study.
* Must agree not to enroll in another study of an investigational agent prior to completion of the study.
* Subjects must be able to understand the requirements of the study and must be accessible and willing to comply with the study procedures even under lock down conditions.
* Ability to provide informed consent.

Phase II (abbreviated):

* Males or females, ages 18 to 85 (inclusive) at the time of screening.
* Negative PCR and no presence of ELISA antibody titers to SARS-CoV-2 at screening.
* Females of childbearing potential and males must be willing to use effective methods of contraception such as hormones (OCP, oral contraceptive pill), condom or occlusive cap with spermicidal agents, intrauterine device (IUD) or intrauterine system (IUS) from at least 14 days prior to vaccination through 90 days following last injection. Male must agree to avoid sperm donation from time of first injection through 90 days following last injection.
* No clinically significant abnormalities in hematology, blood chemistry, or urinalysis laboratory tests at screening.
* Must be willing to forgo blood donation during the blood drawing phase of the study
* Must agree not to enroll in another study of an investigational agent prior to completion of the study.
* Normal oral temperature, pulse rate no greater than 100 beats per minute (sinus rhythm) and controlled blood pressure (in the case of hypertensives under treatment, below 140/90 mmHg).
* Subjects must be able to understand the requirements of the study and must be accessible and willing to comply with the study procedures even under lock down conditions.
* Ability to provide informed consent.

Exclusion Criteria:

Phase I (abbreviated):

* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions or known allergy to the components of the vaccine, including allergy to rice.
* Receipt of investigational product up to 30 days prior to screening or ongoing participation in another clinical trial
* Receipt of licensed vaccines within 14 days of planned study immunization and any AE's possibly related to licensed vaccine immunization at Day 0.
* Inability to observe possible local reactions at the injection sites due to a physical condition or permanent body art.
* Known hemoglobinopathy or coagulation abnormality.
* New onset of fever >37.8 ºC AND [cough OR shortness of breath OR anosmia/ageusia] or any other inter current illness within 14 days prior to screening
* High risk of exposure to SARS-CoV-2 prior to enrollment (close contact, self-isolation at present due to household contact, frontline healthcare provider in contact with COVID-19 subjects).
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health, per the best clinical judgement of the investigator.
* Women who are pregnant or breastfeeding.
* Positive urine pregnancy test or women have an intention to be pregnant during the study.
* Confirmed or suspected illness caused by coronaviruses, SARS-CoV 1, and Middle East Respiratory Syndrome (MERS)-CoV.
* Received any prior vaccine against a coronavirus
* Receipt of blood/plasma products or immunoglobulin, from within 60 days before study intervention administration or planned receipt throughout the study.
* History of alcohol or drug abuse per clinical judgement within 5 years prior to study vaccination.
* Participants who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol.
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study.
* Individuals who are living with severely immunocompromised people (e.g. transplant patients, those under active cancer immunosuppressant therapy), pregnant women, lactating women, children under 12 months old, or any other individual that, in the judgment of the investigator, might be at increased risk.

Phase II (abbreviated):

* History of severe local or systemic reactions to any vaccination or a history of severe allergic reactions or known allergy to the components of the vaccine, including allergy to rice.
* Receipt of investigational product (except of confirmed placebo in IIBR20-001 study) up to 30 days prior to screening or ongoing participation in another clinical trial (except of IIBR20-001 trial).
* Receipt of licensed vaccines within 14 days of planned study immunization and any AE's possibly related to licensed vaccine immunization at Day 0.
* Inability to observe possible local reactions at the injection sites due to a physical condition or permanent body art.
* Known hemoglobinopathy or coagulation abnormality (subjects treated by anticoagulation or anti platelets are not excluded).
* New onset of fever >37.8ºC AND [cough OR shortness of breath OR anosmia/ageusia], or any other inter current illness within 14 days prior to screening
* Factors that increase risk to the subject to severe disease per CDC guidance including the following risk factors (in any case of ambiguous grading, decision will be made per investigator's best clinical judgement): Cancer [ongoing malignancy or recently diagnosed malignancy in the last five years, not including non-melanotic skin cancer], Chronic Kidney Disease (eGFR<60 mL/min/1.73 m^2), liver disease (ALT or AST) > 1.5 × ULN; or alkaline phosphatase and direct bilirubin > ULN (total bilirubin may be up to 2 × ULN as long as direct bilirubin is equal to or below the ULN); or PT INR > 1.25), COPD; Immunocompromised state from solid organ transplant; Obesity (BMI≥30kg/m2); Serious heart conditions, such as heart failure, coronary artery disease, or cardiomyopathies; Sickle cell disease; Type 1/2 diabetes mellitus (HbA1C>8.0%, per medical history questioning or records) ); Asthma; Cerebrovascular disease; Cystic fibrosis, uncontrolled hypertension that does not respond to therapy, Pulmonary fibrosis, Thalassemia.
* Anticipating the need for immunosuppressive treatment within the next 6 months.
* Clinically significant (by means of potentially risking the subject or that would be potentially detrimental to the results of the study) medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health or for severe COVID-19, per the investigator.
* Any progressive or severe neurologic condition/disorder, dementia, seizure disorder, or history of Guillian-Barré syndrome.
* Known or suspected impairment of the immune system including rheumatic, connective tissue or vascular disease of autoimmune origin
* Women who are pregnant or breastfeeding.
* Positive urine or serum pregnancy test or women have an intention to be pregnant during the study.
* Clinically significant abnormal CBC results in WBC, hemoglobin, hematocrit, or platelets.
* Clinically significant abnormal urinalysis: RBC, protein, or glucose only.
* Positive serology for: hepatitis B surface antigen, hepatitis C, HIV.
* Known or suspected illness caused by coronaviruses, SARS-CoV 1, and Middle East Respiratory Syndrome (MERS)-CoV..
* Received any prior vaccine against a coronavirus.
* Receipt of blood/plasma products or immunoglobulin, from within 60 days before study intervention administration or planned receipt throughout the study.
* Immunosuppressive medications received within 90 days before screening. (Not including [1] corticosteroid nasal spray for allergic rhinitis; [2] topical corticosteroids for mild, uncomplicated dermatitis; or [3] oral/parenteral corticosteroids given for non-chronic conditions not expected to recur [length of therapy 10 days or less with completion at least 30 days prior to vaccination].)
* History of alcohol or drug abuse per clinical judgement within 5 years prior to study vaccination (excluding cannabis)
* Participants who, in the judgment of the investigator, will be unlikely to comply with the requirements of this protocol.
* Any other significant finding that in the opinion of the investigator would increase the risk of the individual having an adverse outcome from participating in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 843 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Phase I and II - The number, grade and percentage of study participants who experience any study injection-associated AEs or SAEs. | 365 days post last vaccination
  * Solicited events for 7 days after vaccination.
  * Unsolicited events through 28 days after vaccination.
  * SAEs 365 days after last vaccination
  * New Onset Chronic Medical Condition (NOCMC) or Medically Attended AE (MAAE) 365 days after last vaccination.
Phase II - IIBR-100 Immunogenicity by determining neutralizing antibody titers to SARS-CoV-2 | 28 days post last vaccination
  Immunogenicity will be determined by GMT, GMFR, Seroconversion rates of the neutralizing antibody titers to SARS-CoV-2 per group at 28 days following last vaccination (in relation to Day 0-baseline).

SECONDARY OUTCOMES:
Phase I and II - IIBR-100 Immunogenicity as determined by GMT, GMFR, Seroconversion rates of the neutralizing antibody titers to SARS-CoV-2 at baseline (day 0) and throughout the study | 365 days post last vaccination
  Immunogenicity will be evaluated at the following days: 0, 7±2d, 14±2d, 28±4d, 56±5d, 84±4d, 168±14d, 252±14d and 365±14d after the first vaccination for single-dose groups (prime), and at days 0, 14±2d, 28±4d, 35±4d, 42±4d, 56±5d, 84±4d, 112±14d, 196±14d, 280±14d and 393±14d for the prime-boost groups
Phase I and II - IIBR-100 immunogenicity as determined by GMT, GMFR, Seroconversion rates of the binding antibody titers to SARS-CoV-2 at baseline (day 0) and throughout the study | 365 days post last vaccination
  Immunogenicity will be evaluated at the following days: 0, 7±2d, 14±2d, 28±4d, 56±5d, 84±4d, 168±14d, 252±14d and 365±14d after the first vaccination for single-dose groups (prime), and at days 0, 14±2d, 28±4d, 35±4d, 42±4d, 56±5d, 84±4d, 112±14d, 196±14d, 280±14d and 393±14d for the prime-boost groups
Phase I and II - Cellular immunogenicity as assessed by ELISPOT and ELISA. | 365 days post last vaccination
  Cellular immunogenicity will be assessed at the following days: 0, 28±4d, 56±5d, 84±4d, 168±14d and 365±14d for single dose groups and at days 0, 56±5d, 84±4d, 112±14d, 196±14d and 393±14d for the prime-boost groups.

OTHER OUTCOMES:
Phase I and II - Potential efficacy of IIBR-100 vaccine by means of prevention of COVID-19 disease (as defined by FDA Guidance) | 14 days post last vaccination
  Number of virologically confirmed (PCR positive) symptomatic cases of COVID-19, 14 days after having received on or two active vaccine injections
Phase I and II - Potential efficacy of IIBR-100 vaccine by means of prevention of COVID-19 Severe Disease (per FDA Guidance) | 14 days post last vaccination
  Number of virologically confirmed (PCR positive) severe cases of COVID-19, 14 days after having received on or two active vaccine injections
Phase I and II - Potential efficacy of IIBR-100 vaccine by means of serology confirmed infection (seroconversion to non-vaccine antigen) in combination with one or more of the clinical symptoms proposed. | 14 days post last vaccination
  Number of serology confirmed symptomatic cases of COVID-19, 14 days after having received on or two active vaccine injections
Phase I and II - Kinetics evaluation of antibody decline based on temporal sub-group analyses | 365 days
  Kinetics of antibody decline based on temporal sub-group analyses (at 3, 6, 9, 12 months post first vaccination)

CONTACTS AND LOCATIONS:
Locations (8):
- Israel (8):
  - Assuta - University Hospital, Ashdod
  - Barzilai MC, Ashkelon
  - Rambam MC, Haifa
  - Hadassah Medical Center, Jerusalem
  - Meir MC, Kfar Saba
  - Rabin MC, Petah Tikva
  - Sheba Medical Center Hospital- Tel Hashomer, Ramat Gan
  - Sourasky MC, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caraco Y, Madar-Balakirski N, Ben-Ami E, Zeltser D, Maayan S, Eliakim-Raz N, Peer A, Brosh-Nissimov T, Vishlitzky V, Beth-Din A, Bar-Haim E, Israely T, Paran N, Fisher M, Hoggeg M, Atsmon J, Cohen D, Goldstaub D, Levin Y, Danon Y, Panet A, Shapira S, Yitzhaki S, Marcus H. Using the vesicular stomatitis virus vector (rVSV vector) platform for SARS-CoV-2 vaccine development: Phase 1/2 safety and immunogenicity of IIBR-100 in healthy adults. Vaccine. 2025 Nov 20;67:127837. doi: 10.1016/j.vaccine.2025.127837. Epub 2025 Oct 16. PMID 41106035